CLINICAL TRIAL: NCT02613052
Title: The Use of Agitated Saline, Albumin, or a Propofol-albumin Mixture for Enhanced Contrast in Bubble Studies During Transesophageal Echocardiographic Examinations
Brief Title: Agitated Saline, Albumin, or Propofol-albumin Mixture for Enhanced Contrast in TEE Examinations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Swapnil Khoche, Assistand Clinical Professor, University of California, San Diego
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Diagnostic
Other Study IDs: 151360
Record Dates: First submitted 2015-11-19; First posted 2015-11-24 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Transesophageal Echocardiography Contrast Agents
MeSH Terms: interventions — Saline Solution; Sodium Chloride; Serum Albumin, Human; Propofol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Agitated Normal Saline (Placebo Comparator): Agitated saline is the current standard of care contrast agent used for bubble studies. 10 mL of agitated normal saline will be used for the bubble study.
  Interventions: Drug: normal saline
- Albumin only (Active Comparator): 10 mL of agitated 5% albumin will be used for the bubbly study.
  Interventions: Drug: human albumin
- Albumin and Propofol (Experimental): 7 mL of 5% albumin and 3 mL of propofol (10 mg/mL) will be agitated together and used for the bubble study.
  Interventions: Drug: human albumin and propofol

INTERVENTIONS:
Drug: normal saline — 10 mL of normal saline agitated prior to IV administration
  Other Names: sodium chloride
  Arms: Agitated Normal Saline
Drug: human albumin — 10 mL of 5% albumin agitated prior to IV administration
  Arms: Albumin only
Drug: human albumin and propofol — 7 mL of 5% albumin mixed with 3 mL of propofol (10 mg/mL) agitated together prior to IV administration
  Other Names: Diprivan
  Arms: Albumin and Propofol

SUMMARY:
This is a prospective, randomized, controlled study to determine if albumin and propofol or albumin only will provide superior qualitative contrast enhancement during TEE bubble studies compared to agitated saline. Each patient will receive three randomized bubble studies (agitated saline, albumin, and albumin and propofol) using 10 ml of agitated contrast agent. The albumin and propofol mixture will consist of 7 mL of 5% albumin plus 3 mL of propofol (10 mg/mL). Each patient will undergo qualitative review of all 3 bubble studies by 10 different anesthesiologists and/or cardiologists credentialed to read echocardiographic studies at the time of the surgical procedure, and also with retrospective review of the echo video (~200 studies). A bicaval view will be obtained to record a 20 beat loop for each bubble study. Hemodynamic variables prior to injection of contrast agent; and 30 seconds, 1 minute and 2 minutes after injection will be monitored and recorded.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled study to determine if albumin and propofol or albumin only will provide superior qualitative contrast enhancement during TEE bubble studies compared to the current standard of care contrast agent, agitated saline. The study will take place in the Operating Rooms (OR) at the UCSD Sulpizio Cardiovascular Center. The TEE studies will be reviewed by UCSD Anesthesiology or Cardiology faculty who are credentialed to read and interpret echocardiographic studies.

The study population will consist of 20 English-speaking patients and all will receive two doses of contrast, namely agitated albumin or propofol and albumin mixture, undergoing cardiac surgery who require TEE. Each patient will undergo qualitative review by 10 anesthesiologists and/or cardiologists credentialed to read echocardiographic studies at the time of the surgical procedure, and also with retrospective review of the echo video. The multiple reviewers per patient will increase the power of the study (~200 studies). Each patient will receive three bubble studies using 10 ml of agitated contrast agent as named above. The order in which each contrast agent is utilized, as well as the experimental contrast agent, is randomized and the interpreting physician is blinded to this information. Agitated saline (AS) alone will be used as a (third dose) control for each patient, which is the current standard contrast agent for TEE bubble studies. The other bubble studies will use an experimental agitated contrast agent, either a mixture of 7 mL albumin and 3 mL propofol (10 mg/ml) or 10 mL albumin (human). Saline and albumin 5% are intravenous fluids FDA approved for the use in restoration and maintenance of circulating of blood volume. Propofol is FDA approved for the use in induction or maintenance of general anesthesia.

The anesthesia care team, as per the standard care during UCSD cardiac surgical procedures, will place a TEE probe after induction of general anesthesia and endotracheal intubation. During the initial TEE exam, a bicaval view will be obtained. Both the order and type of experimental agitated contrast agent will be randomized and blinded to the sonographer and reviewer. A 20 beat loop will be recorded for each bubble study. Hemodynamic variables prior to injection of contrast agent; and 30 seconds, 1 minute and 2 minutes after injection are monitored and recorded. All recorded data will be anonymized prior to review. TEE is standard of care and routinely used in the care of cardiac surgery patients and is not performed solely for this study.

All anesthetic, surgical and medical interventions will be chosen and carried out by the surgical and anesthesia teams, including those involving invasive monitor placement, fluid administration, ventilator management and patient positioning.

Appropriate statistical analysis will be utilized to evaluate the difference in contrast enhancement in the saline only, albumin, and albumin and propofol groups.

The results of the study will be published in the peer-reviewed medical literature.

ELIGIBILITY:
Inclusion Criteria:

* cardiac surgical patients requiring a transesophageal echocardiogram (TEE)

Exclusion Criteria:

* allergy to propofol
* inability to place a TEE probe
* inability to obtain a TEE bicaval image
* known right to left intracardiac shunt
* pt refusal to accept human blood products including albumin
* pt refusal to participate in study
* vulnerable patients (pregnant women, prisoners, cognitively impaired, or institutionalized)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Qualitative enhancement in right atrial opacification during intraoperative TEE bubble studies | 6 months
  Number of participants with qualitatively enhanced right atrial opacification with albumin or albumin and propofol mixture compared to standard of care agitated normal saline, during TEE bubble studies using the bicaval view.

CONTACTS AND LOCATIONS:
Overall Officials: Swapnil Khoche, MD, Principal Investigator — University of California, San Diego; Ryan YS Suda, MD, Study Director — University of California, San Diego
Locations (1):
- UC San Diego Sulpizio Cardiovascular Center, La Jolla, California, United States

REFERENCES:
- [Background] Meerbaum S. Introduction and general background. In: Myocardial Contrast Two-Dimensional Echocardiography, Meerbaum S, Meltzer R (Eds), Kluwer Academic Publishers, Boston 1989. p.2
- [Background] Stewart MJ. Contrast echocardiography. Heart. 2003 Mar;89(3):342-8. doi: 10.1136/heart.89.3.342. No abstract available. PMID 12591856
- [Background] Attaran RR, Ata I, Kudithipudi V, Foster L, Sorrell VL. Protocol for optimal detection and exclusion of a patent foramen ovale using transthoracic echocardiography with agitated saline microbubbles. Echocardiography. 2006 Aug;23(7):616-22. doi: 10.1111/j.1540-8175.2006.00272.x. PMID 16911341
- [Background] Unger EC, Porter T, Culp W, Labell R, Matsunaga T, Zutshi R. Therapeutic applications of lipid-coated microbubbles. Adv Drug Deliv Rev. 2004 May 7;56(9):1291-314. doi: 10.1016/j.addr.2003.12.006. PMID 15109770
- [Background] Mulvagh SL, Rakowski H, Vannan MA, Abdelmoneim SS, Becher H, Bierig SM, Burns PN, Castello R, Coon PD, Hagen ME, Jollis JG, Kimball TR, Kitzman DW, Kronzon I, Labovitz AJ, Lang RM, Mathew J, Moir WS, Nagueh SF, Pearlman AS, Perez JE, Porter TR, Rosenbloom J, Strachan GM, Thanigaraj S, Wei K, Woo A, Yu EH, Zoghbi WA; American Society of Echocardiography. American Society of Echocardiography Consensus Statement on the Clinical Applications of Ultrasonic Contrast Agents in Echocardiography. J Am Soc Echocardiogr. 2008 Nov;21(11):1179-201; quiz 1281. doi: 10.1016/j.echo.2008.09.009. PMID 18992671
- [Background] Porter TR, Abdelmoneim S, Belcik JT, McCulloch ML, Mulvagh SL, Olson JJ, Porcelli C, Tsutsui JM, Wei K. Guidelines for the cardiac sonographer in the performance of contrast echocardiography: a focused update from the American Society of Echocardiography. J Am Soc Echocardiogr. 2014 Aug;27(8):797-810. doi: 10.1016/j.echo.2014.05.011. No abstract available. PMID 25085408
- [Background] Shapiro JR, Reisner SA, Lichtenberg GS, Meltzer RS. Intravenous contrast echocardiography with use of sonicated albumin in humans: systolic disappearance of left ventricular contrast after transpulmonary transmission. J Am Coll Cardiol. 1990 Dec;16(7):1603-7. doi: 10.1016/0735-1097(90)90308-c. PMID 2254545
- [Background] Davison P, Clift PF, Steeds RP. The role of echocardiography in diagnosis, monitoring closure and post-procedural assessment of patent foramen ovale. Eur J Echocardiogr. 2010 Dec;11(10):i27-34. doi: 10.1093/ejechocard/jeq120. PMID 21078836
- [Background] Baker MT, Naguib M. Propofol: the challenges of formulation. Anesthesiology. 2005 Oct;103(4):860-76. doi: 10.1097/00000542-200510000-00026. PMID 16192780
- [Background] de Jong N, Emmer M, van Wamel A, Versluis M. Ultrasonic characterization of ultrasound contrast agents. Med Biol Eng Comput. 2009 Aug;47(8):861-73. doi: 10.1007/s11517-009-0497-1. Epub 2009 May 26. PMID 19468770
- [Background] Kitzman DW, Goldman ME, Gillam LD, Cohen JL, Aurigemma GP, Gottdiener JS. Efficacy and safety of the novel ultrasound contrast agent perflutren (definity) in patients with suboptimal baseline left ventricular echocardiographic images. Am J Cardiol. 2000 Sep 15;86(6):669-74. doi: 10.1016/s0002-9149(00)01050-x. PMID 10980221
- [Background] Dewhirst E, et al. The Use of a Propofol-Saline Mixture for Enhanced Contrast in Bubble Studies During Echocardiographic Examinations. Society of Pediatric Anesthesia Meeting (Winter 2012).
- [Background] Geny B, Mettauer B, Muan B, Bischoff P, Epailly E, Piquard F, Eisenmann B, Haberey P. Safety and efficacy of a new transpulmonary echo contrast agent in echocardiographic studies in patients. J Am Coll Cardiol. 1993 Oct;22(4):1193-8. doi: 10.1016/0735-1097(93)90437-6. PMID 8409060